CLINICAL TRIAL: NCT03050632
Title: An Investigation of the Effects of Cognitive and Emotional Functioning on Treatment Outcomes
Brief Title: Effects of Cognitive and Emotional Functioning on Treatment Outcomes
Acronym: CEO
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: With change of personnel and lab resources, this study was not feasible without independent funding
Sponsor: Boston University Charles River Campus (Other)
Responsible Party: Principal Investigator, Michael Otto, Professor of Psychology, Boston University Charles River Campus
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 4209
Record Dates: First submitted 2017-01-02; First posted 2017-02-13 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Eating Disorders
Keywords: working memory; adherence
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Working Memory Intervention (N-back) (Experimental): Participants will complete the working memory priming task either for the first 3 days of the intervention or the last 3 days of the intervention, with order counterbalanced across participants. The working memory prime is the N-back test, a measure of working memory in which individuals need to make a response to targets which are repeated letters either in a row (i.e., one-back) or in every-other-letter format (i.e., two-back) (Jaeggi et al., 2010).
  Interventions: Behavioral: N-back
- "White Bear" Task (Placebo Comparator): Participants will complete this non-working-memory control task either for the first 3 days of the intervention or the last 3 days of the intervention, depending on counterbalanced order. The task consists of a procedure developed by Wegner and colleagues (1987) in a study of thought suppression, which instructs participants to inhibit thoughts of a white bear, and to indicate with a pencil mark every time the thought of the white bear occurs to them.
  Interventions: Behavioral: White Bear Task

INTERVENTIONS:
Behavioral: N-back — The N-back task is a measure of working memory in which individuals need to make a response to targets which are repeated letters either in a row (i.e., one-back) or in every-other-letter format (i.e., two-back).
  Arms: Working Memory Intervention (N-back)
Behavioral: White Bear Task — For this thought suppression task, participants are instructed to inhibit thoughts of a white bear, and to indicate with a pencil mark every time the thought of the white bear occurs to them.
  Arms: "White Bear" Task

SUMMARY:
The investigators are interested about the degree to which individuals can persist with individualized treatment goals when their cues (external such as food, or internal such as anxiety) are high for impulsive/maladaptive behavior (e.g., purging, not eating, etc.). The investigators want to find specific high-difficulty situations in which to assess whether participants remain mindful of the big picture and are willing to work toward therapeutic goals. Also, the investigators want to rate the participants degree of success (e.g., proportion of calories eaten) assessed more objectively.

The theory is that working memory capacity (WMC) modulates the ability to keep longer-term goals in mind when faced by current stress/temptations. For example, the ability to control drinking when one has an implicit urge to drink is predicted by WMC. The ability to apply a novel emotional regulation skill at a time of stress is also predicted by WMC. Indeed, the generic ability to pursue goals in the future (as assessed by the discounting of the value of future goals) is reliably predicted by WMC. There is also evidence that activation of brain regions associated with WMC (by direct activation of the dorsolateral prefrontal cortex via transcranial magnetic stimulation (TMS), or by having a person complete a relevant cognitive task) improves delay discounting.

Accordingly, the investigators are proposing a study that both assesses the link between WMC and relevant the clinical measures noted above, as well as changes in these measures following activation of WM with a cognitive prime (WM task). The overall design calls for an initial WMC assessment, followed by randomization to complete 3 days of a WM prime and then 3 days of a no prime group, or vice versa. The investigators then assess the clinical outcomes noted above across the following 6 days, with a WM prime first or no prime first occurring prior to the targeted behaviors. The investigators will prime WM prior to participant's evening meal, with the WM intervention offered during the free time before this meal.

ELIGIBILITY:
Inclusion Criteria:

* Residential patients
* Females 18 and older
* Able to provide informed consent for the study
* Sufficient command of the English language
* Have experience using a computer and mouse
* Diagnosed with an Eating Disorder

Exclusion Criteria:

None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Meal Compliance | Comparison of day 5 to day 8 scores taking into account intervention type, intervention order, and baseline scores
  Therapeutic Food and Snack Log.

SECONDARY OUTCOMES:
Mood | Comparison of day 5 to day 8 scores taking into account intervention type, intervention order, and baseline scores
  Mood Monitoring Form
Delay Discounting | Comparison of day 5 to day 8 scores taking into account intervention type, intervention order, and baseline scores
  Monetary-Choice Questionnaire
Eating Disorder Symptoms | Comparison of day 5 to day 8 scores taking into account intervention type, intervention order, and baseline scores
  Eating Disorder Diagnostic Scale (EDDS)
Depression | Comparison of day 5 to day 8 scores taking into account intervention type, intervention order, and baseline scores
  Center for Epidemiologic Studies Depression Scale (CES-D)
Depression, Anxiety, and Stress | Comparison of day 5 to day 8 scores taking into account intervention type, intervention order, and baseline scores
  Depression Anxiety Stress Scales (DASS-21)

CONTACTS AND LOCATIONS:
Locations (1):
- Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No